CLINICAL TRIAL: NCT05380466
Title: The Effect of "Quantum Touch" Application on Transfer Anxiety in Pediatric Patients and Their Parents Planned to Be Hospitalized in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Eda Polat, Research Assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IstanbulMU16
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anxiety; Child, Only; Emergencies
MeSH Terms: conditions — Anxiety Disorders; Emergencies

STUDY DESIGN:
Intervention Model Description: Parallel group, randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quantum Touch (Experimental): Those who are planned to be hospitalized from the emergency department and applied quantum touch
  Interventions: Other: Quantum Touch
- Control (No Intervention): Those who are planned to be hospitalized from the emergency department and who have not intervention

INTERVENTIONS:
Other: Quantum Touch — Quantum-Touch is one of the therapeutic touch techniques, a biofield therapy that uses life force energy to facilitate healing
  Arms: Quantum Touch

SUMMARY:
Anxiety, which is a subjective experience in which many emotions such as worry, uncertainty, restlessness, and sadness are experienced together, is defined as "a state of tension that arises as a result of the internal conflict experienced by the individual". Emergency services are the units where all kinds of patients and injured are followed and treated 24 hours a day, and anxiety is a very common emotional reaction in patients who apply to the emergency department and their relatives. The patient and his family; They experience varying levels of anxiety due to a sudden and unexpected deterioration of health, the threat of their life, the uncertainty of the situation, the fear of death, role changes, disruption of routines, and being in an unfamiliar hospital environment. With the increase of anxiety, distraction in family members, repetitive questions to health personnel, inability to understand the importance of the event and difficulty in making decisions can be seen.Leaving the emergency room as well as being in the emergency room causes anxiety in individuals. The anxiety experienced in this situation is called transfer anxiety. Transfer anxiety is often defined as "anxiety experienced by an individual when he/she moves from a safe and familiar environment to an unfamiliar environment" and was accepted as a nursing diagnosis by NANDA in 1992. Transferring the patient from the emergency room to the clinic is a routine procedure for emergency nurses, but it causes anxiety for the patient and their relatives. As a result of transfer anxiety, many patients and their family members experience widespread confusion both before and after transfer and tend to certain problems. The patient and family members experience anxiety when they are in a foreign environment with different routines and follow-up procedures for the first time and do not know what to expect. Pharmacological and non-pharmacological methods are used to reduce anxiety. Cognitive behavioral therapy techniques are frequently used among non-pharmacological methods. Cognitive-behavioral therapies are a form of treatment developed on the basis of behavioral psychological counseling theory, which is problem-focused, deals with the "here and now" and applies learning theories to help individuals when they encounter difficulties and life problems that they cannot overcome in their daily lives. Cognitive-behavioral therapies that are highly suitable for working with children, youth, adults, the elderly and families; They are easy to work with individually or in groups and do not require any hardware. Among cognitive behavioral therapy techniques, therapy strategies that reduce anxiety include relaxation, biofeedback, systematic desensitization, exercise, vestibular desensitization, response prevention, and therapeutic touch techniques. Therapeutic touch; In 1972, it was started to be used as a healing method by the manipulation of hypothetical human bioenergy field by nurse professor Doores Krieger. In the literature, it is frequently applied to reduce pain and anxiety in nursing studies and successful results are obtained. Quantum-Touch; It is one of the therapeutic touch techniques and is a biofield therapy that uses life force energy to facilitate healing. Quantum-Touch was first described by Richard Gordon and Bob Rasmusson in 1978; It activates life force energy by combining various hand positions, various breathing techniques and body awareness exercises. It is applied by directing the formed high energy field to an area of pain, stress or illness through therapeutic touch. Tully (2017) found that Quantum Touch in reducing acute and chronic pain; Walton (2011) reported that Quantum-Touch application is effective in chronic musculoskeletal pain. The patient and/or the patient's family may be physically ready for relocation in the hospital environment, but they are not psychologically ready. Inadequate preparation of the individual for the transfer from the emergency room to the clinic or lack of information about the transfer, perceiving that his safety is under threat, and experiencing uncertainty about his situation cause transfer anxiety. Although it is seen in the literature that transfer anxiety is applied in adults and generally in intensive care units, no study has been found in children and emergency services.

DETAILED DESCRIPTION:
Anxiety, which is a subjective experience in which many emotions such as worry, uncertainty, restlessness, and sadness are experienced together, is defined as "a state of tension that arises as a result of the internal conflict experienced by the individual". Emergency services are the units where all kinds of patients and injured are followed and treated 24 hours a day, and anxiety is a very common emotional reaction in patients who apply to the emergency department and their relatives. The patient and his family; They experience varying levels of anxiety due to a sudden and unexpected deterioration of health, the threat of their life, the uncertainty of the situation, the fear of death, role changes, disruption of routines, and being in an unfamiliar hospital environment. With the increase of anxiety, distraction in family members, repetitive questions to health personnel, inability to understand the importance of the event and difficulty in making decisions can be seen.Leaving the emergency room as well as being in the emergency room causes anxiety in individuals. The anxiety experienced in this situation is called transfer anxiety. Transfer anxiety is often defined as "anxiety experienced by an individual when he/she moves from a safe and familiar environment to an unfamiliar environment" and was accepted as a nursing diagnosis by NANDA in 1992. Transferring the patient from the emergency room to the clinic is a routine procedure for emergency nurses, but it causes anxiety for the patient and their relatives. As a result of transfer anxiety, many patients and their family members experience widespread confusion both before and after transfer and tend to certain problems. The patient and family members experience anxiety when they are in a foreign environment with different routines and follow-up procedures for the first time and do not know what to expect. Pharmacological and non-pharmacological methods are used to reduce anxiety. Cognitive behavioral therapy techniques are frequently used among non-pharmacological methods. Cognitive-behavioral therapies are a form of treatment developed on the basis of behavioral psychological counseling theory, which is problem-focused, deals with the "here and now" and applies learning theories to help individuals when they encounter difficulties and life problems that they cannot overcome in their daily lives. Cognitive-behavioral therapies that are highly suitable for working with children, youth, adults, the elderly and families; They are easy to work with individually or in groups and do not require any hardware. Among cognitive behavioral therapy techniques, therapy strategies that reduce anxiety include relaxation, biofeedback, systematic desensitization, exercise, vestibular desensitization, response prevention, and therapeutic touch techniques. Therapeutic touch; In 1972, it was started to be used as a healing method by the manipulation of hypothetical human bioenergy field by nurse professor Doores Krieger. In the literature, it is frequently applied to reduce pain and anxiety in nursing studies and successful results are obtained. Quantum-Touch; It is one of the therapeutic touch techniques and is a biofield therapy that uses life force energy to facilitate healing. Quantum-Touch was first described by Richard Gordon and Bob Rasmusson in 1978; It activates life force energy by combining various hand positions, various breathing techniques and body awareness exercises. It is applied by directing the formed high energy field to an area of pain, stress or illness through therapeutic touch. Tully (2017) found that Quantum Touch in reducing acute and chronic pain; Walton (2011) reported that Quantum-Touch application is effective in chronic musculoskeletal pain. The patient and/or the patient's family may be physically ready for relocation in the hospital environment, but they are not psychologically ready. Inadequate preparation of the individual for the transfer from the emergency room to the clinic or lack of information about the transfer, perceiving that his safety is under threat, and experiencing uncertainty about his situation cause transfer anxiety. Although it is seen in the literature that transfer anxiety is applied in adults and generally in intensive care units, no study has been found in children and emergency services.

ELIGIBILITY:
Inclusion Criteria:

* Being between 5-10 years old (the fear scale used for children can be used for 5-10 years old)
* Planning hospitalization from the emergency department to the clinic
* Absence of any mental and/or physical health problems that would prevent communication
* Parents and children speak Turkish
* Parent and child volunteer to participate in the study.

Exclusion Criteria:

Being under 5 years old and over 10 years old

* Having any mental and/or physical health problems that prevent communication
* Parents and children do not agree to participate in the study.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Child Fear Scale | 6 months
  The CFS is a scale from 0 to 4, consisting of five drawn facial expressions ranging from neutral (0=no anxiety) to frightened face (4=severe anxiety).
Child Anxiety Scale-State | 6 months
  CAS-S is similar to a thermometer with a light bulb at the bottom and horizontal lines at intervals that go up. The scale is aimed at children between the ages of four and ten. To measure state anxiety (CAS-S), the child is asked to mark what he feels "right now".

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Zeynep Kamil Gynecology and Pediatrics Training and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The authors will decide and plan among themselves.

REFERENCES:
- [Background] Alp FY, Yucel SC. The Effect of Therapeutic Touch on the Comfort and Anxiety of Nursing Home Residents. J Relig Health. 2021 Jun;60(3):2037-2050. doi: 10.1007/s10943-020-01025-4. PMID 32415423
- [Background] Busch M, Visser A, Eybrechts M, van Komen R, Oen I, Olff M, Dokter J, Boxma H. The implementation and evaluation of therapeutic touch in burn patients: an instructive experience of conducting a scientific study within a non-academic nursing setting. Patient Educ Couns. 2012 Dec;89(3):439-46. doi: 10.1016/j.pec.2012.08.012. Epub 2012 Sep 17. PMID 22995597
- [Background] Ersig AL, Kleiber C, McCarthy AM, Hanrahan K. Validation of a clinically useful measure of children's state anxiety before medical procedures. J Spec Pediatr Nurs. 2013 Oct;18(4):311-9. doi: 10.1111/jspn.12042. Epub 2013 Jun 25. PMID 24094126
- [Background] McKinley S, Coote K, Stein-Parbury J. Development and testing of a Faces Scale for the assessment of anxiety in critically ill patients. J Adv Nurs. 2003 Jan;41(1):73-9. doi: 10.1046/j.1365-2648.2003.02508.x. PMID 12519290
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Senderovich H, Ip ML, Berall A, Karuza J, Gordon M, Binns M, Wignarajah S, Grossman D, Dunal L. Therapeutic Touch((R)) in a geriatric Palliative Care Unit - A retrospective review. Complement Ther Clin Pract. 2016 Aug;24:134-8. doi: 10.1016/j.ctcp.2016.06.002. Epub 2016 Jun 21. PMID 27502814
- [Background] Yucel SC, Arslan GG, Bagci H. Effects of Hand Massage and Therapeutic Touch on Comfort and Anxiety Living in a Nursing Home in Turkey: A Randomized Controlled Trial. J Relig Health. 2020 Feb;59(1):351-364. doi: 10.1007/s10943-019-00813-x. PMID 30982141
- [Background] Zolfaghari M, Eybpoosh S, Hazrati M. Effects of therapeutic touch on anxiety, vital signs, and cardiac dysrhythmia in a sample of Iranian women undergoing cardiac catheterization: a quasi-experimental study. J Holist Nurs. 2012 Dec;30(4):225-34. doi: 10.1177/0898010112453325. Epub 2012 Jul 24. PMID 22828950